CLINICAL TRIAL: NCT03636386
Title: Effectiveness of Percutaneous Microelectrolysis in the Decrease of Pain in Myofascial Trigger Points: Evaluation Through Algometry and Visual Analog Scale. Randomized Controlled Trial.
Brief Title: Percutaneous Microelectrolysis on Myofascial Trigger Points Pain.
Acronym: MEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quiropraxia y Equilibrio (Other)
Collaborators: Universidad Nacional Andres Bello (Other)
Responsible Party: Principal Investigator, Hernán Andrés de la Barra Ortiz, Clinical Professor, Quiropraxia y Equilibrio
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 60312069
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Results first posted 2020-04-15 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Myofascial Trigger Point Pain (MTrP)
Keywords: Electrotherapy; Electrolysis; Myofascial pain syndromes; Pain Threshold; Analogue visual scale
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Ultrasonic Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous microelectrolysis group (MEP) (Experimental): Group exposed to direct current application using an acupuncture needle with intensities in microamps (μA) in MTrP of upper trapezius muscle. Acupuncture needle correspond to negative electrode or cathode. This group was also be treated with conventional ultrasound (US) before MEP application. US treatments parameters will include; 1MHz, 1.5W/cm2, 5cm2 ERA, 100% duty cycle and 15 minutes treatment time.
  Interventions: Device: Percutaneous microelectrolysis; Device: Ultrasound therapy
- Ultrasound therapy (Active Comparator): Group treated with conventional ultrasound (US) on MTrP with 1MHz, 1.5W/cm2, 5cm2 ERA, 100% duty cycle and 15 minutes treatment time.
  Interventions: Device: Ultrasound therapy

INTERVENTIONS:
Device: Percutaneous microelectrolysis — 284/5000 Application of Direct Current through an acupuncture needle with intensities in microamps (μA) in the PGm of the upper trapezius muscle. The acupuncture needle will correspond to the negative electrode or cathode. The intensity of work will be 610μA at the myofascial trigger point.
  Other Names: Electrolysis through the polar effect of the cathode
  Arms: Percutaneous microelectrolysis group (MEP)
Device: Ultrasound therapy — Application of conventional ultrasound (US) on PGm with a frequency of treatment 1MHz, intensity of 1.5W / cm2, ERA 5cm2, Duty Cycle 100%, treatment time 6 minutes.
  Other Names: Treatment with conventional ultrasound

SUMMARY:
The aim of the design is to investigate the value of percutaneous microelectrolysis (MEP) as an analgesic technique in myofascial trigger points. This research seeks to evaluate influence of cathode polar effects on the reduction of painful pressure (PPT) threshold and pain intensity (PI) in the myofascial trigger points (MTrPs) of upper trapezius muscle. An assessment with algometry and visual analog scale (VAS) will be made before applying the intervention. The study will evaluate changes in PPT and PI in a group exposed to percutaneous microelectrolysis (MEP) aplication compared to control group. Both groups will be provided with a baseline treatment of therapeutic ultrasound. Treatment will include three evaluation sessions. Subsequently, researchers will proceed to compare PPT and PI obtained from algometry test and VAS in each groups, and between groups, before and after the intervention. Changes obtained between sessions will be compared.

DETAILED DESCRIPTION:
1. Methodological design

   Type: Experimental, randomized clinical trial (RCT).

   1.1 Study population. Students of Science Rehabilitation Faculty (SRF) of Andrés Bello University constituted by the careers of Kinesiology, Occupational Therapy and Speech Therapy.

   1.2 Ethical aspects of research. Study was approved by ethics committee of Metropolitan East Health Service (SSMO),Santiago de Chile, to ensure compliance with bioethical regulations. Study was approved by Bioethics Committee on June 26, 2018. An informed consent will be applied to participants in which the study and intervention procedures will be explained.
2. Variables. 2.1 Conceptual definition of the variables • Pain pressure threshold (PPT): magnitude of pain in Kg/cm2 reported by participants when performing algometry test in upper trapezius muscle.

   * Pain Intensity (PI): magnitude of pain in millimeters (mm) referred by participants when performing the pressure algometry test in MTrP of upper trapezius muscle.
   * Percutaneous Microelectrolysis (MEP): application of direct current through an acupuncture needle with intensities in microamps (μA) in the MTrP of upper trapezius muscle. Acupuncture needle will correspond to negative electrode or cathode. Intensity will be 610μA at MTrP.
   * Therapeutic ultrasound: conventional ultrasound application (US) on MTrP with a 1MHz treatment frequency, 1.5W/cm2, 5cm2 ERA, 100% duty cycle, 15 minutes treatment time. US therapy was applied to both groups equally as baseline traetment.

   2.2 Operational definition of the variables

   • Pain pressure threshold (PPT): pressure trough algometry in MTrPs of upper trapezius muscle. UPD values will be recorded in Kg/cm2. PPT will be evaluated through the BASELINE® pressure algometer.

   • Pain Intensity: Evaluated through Visual Analogue Scale (VAS) at moment of performing pressure algometry in MTrPs of upper trapezius muscle.

   2.3 Type of variable definition

   • Pain pressure threshold (PPT): Dependent, quantitative, reason variable.

   • Pain intensity (ID): Dependent, quantitative, interval variable.

   • Percutaneous Microelectrolysis (MEP): independent, quantitative, interval variable.

   • Therapeutic ultrasound: independent variable, quantitative, reason.

   3.1 Investigation place Study will be conducted at the physioterapy laboratory of SRF, building C5 room 401 of Andrés Bello University, Avenue Fernández Concha 700, Las Condes.

   3.2 Inclusion criteria

   - Participants over 18 years old.

   - Students of SRF.

   - Positive hypersensitive MTrPs. A PPT less than 3Kg/cm2 was considered as positive MTrP.

   3.3 Exclusion criteria
   * Neck or shoulders pathologies in the last 6 months (as fractures, sprains, tendinopathies, dislocations or muscle tears).
   * Cervical pain, sensitivity alterations such as hyposthesia, anesthesia or hyperesthesia in neck, shoulders and/or arms.
   * Wounds or skin alterations in shoulder as psoriasis, scars or keloids.
   * Fear to electrotherapy application.
   * Analgesic pharmacological treatment at recruitment time (non-steroidal anti-inflammatory or steroidal drugs).

   3.4 Elimination Criteria
   * Non-tolerance electrotherapy intervention
   * Non-completion of evaluation protocol

4. Material and Methods Present design represents a randomized double-blind clinical trial. Study was approved on June 18, 2019 by Eastern Metropolitan Health Service of Santiago (SSMO) ethics committee. Study was registered at www.clinicaltrials.gov. Participants were divided in two groups assessed in both presences of MTrPS in shorter upper trapezius muscle. It was recording the PPT and PI before and after intervention. Both groups received therapeutic ultrasound as baseline treatment. Experimental group received microelectrolysis additionally. A reassessment of PPT and PI was done on day one, three and seven post intervention.

Subjects. forty-eight healthy volunteers were recruited (23 men, 25 women, average age 22 years). Participants were students of Science Rehabilitation Faculty (SRF) of Andrés Bello University, Santiago de Chile. Number of participants was selected by convenience. An invitation was extended to students through formal communication channels (mailing), student representatives and social networks, summoning two hundred and seven potential participants. Selection was based on a survey whose first part was structured in relation to general demographic participant's data, including name, age, sex, body mass index (BMI), career year, and personal information contact (e-mail and cell phone number). Second part of survey consisted of closed questions constructed by eligibility criteria. Secondary variables as short upper trapezius muscle laterality (SUTL) and sex were represented as frequencies, while MTrP location distance (MLD) and age was represented as median and BMI in averages. Primary variables included PPT and PI pre-intervention (PPTpre and PIpre) were expressed as averages with their corresponding standard deviation (x, SD). Data were analyzed to compare homogeneity of groups with STATAv.13 program.

Equipment. GYMNA´s COMBI 500 electric stimulator was used for ultrasound application at 1MHz, 1.5Watts/cm2, 100% duty cycle, 5cm2 ERA and 15 minutes.24 SVELTIA´s DC equipment was used for MEP application. It was used a dispersing electrode (area 28.26cm2) and an acupuncture needle (0.3x25millimeters). Circuit was closed by placing dispersing electrode in contralateral arm to trapezius muscle to be treated. Current intensity was 600µA at the needle (current density of 1.71mA/cm2).

Measurement tools. BASELINE® pressure algometer was used to measure PPT (1cm2 surface area).25 Algometry was applied after shortness upper trapezius assessment by placing algometer at the MTrP exerting a perpendicular pressure until user reported pain. Kilograms of pressure per square centimeter (Kg/cm2) was registered. PI was evaluated with VAS. VAS was applied after algometry recording pain perceived with algometry test.

Procedure.

1. Participants 207 surveys were analyzed obtaining 59 potential participants, dropping out five. 54 participants agreed to participate and gave their written consent. Six participants were excluded due absence of MTrPS, obtaining 48 participants (23 men, 25 women). Principal investigator assigned a number to each participant to perform randomization. Conformation of groups was carried out by simple randomization by dark envelopes. Participants didn´t know assigned group and were individually cited in following two weeks to physiotherapy laboratory of SRF to be evaluated.
2. Groups. Sample was divided by a simple randomization process performed with a random number table, assigned participants to one of two study groups. Sequence of randomization and participants of each group was only known by principal investigator. Working groups were designated as experimental (MEP group, n = 24) and control group (n = 24). None subjects knew the treatment that would be applied. Each participant was evaluated registering their age, BMI and SUTL. Location of MTrP was determined at shortness trapezius muscle, taking as reference a line between superior acromion´s midpoint surface and C7 spinous process (PE-AC distance). Algometry and VAS was subsequently applied obtaining the PPT and PI pre intervention (PPTpre y PIpre). Variables described were compared between groups to assess the homogeneity of them. Data obtained reflect the homogeneity of groups at the beginning of the study.
3. Pain pressure threshold (PPTpre) and pain intensity (PIpre) preintervention evaluation.

   A blinded physiotherapist registered PPT and PI before and after participant's intervention. Evaluation station consisted of a chair and a table with the algometer and VAS. The subjects sat with their backs supported with both feet on the floor. Evaluator proceeded to measure both upper trapezius muscles length manually, choosing the shortest. Subsequently a line was drawn between C7 spinous process and upper acromion midpoint face of ipsilateral shoulder. Most sensitive palpation´s point was searched on the line and then marked with a cross measuring distance from C7 to this point. Algometry was applied at selected point exerting a perpendicular pressure until the user referred pain. Participants were instructed to raise slightly contralateral hand when feeling pain in algometry test. A PPT less than 3Kg/cm2 was recorded as a positive MTrP. This was same protocol used for participants pre-selection where 6 of 54 were excluded. Next pain intensity was assessed with VAS, recording pain magnitude in millimeters produced by algometry. PPTpre and PIpre data were tabulated in Microsoft excel® program sheet.
4. Therapeutic ultrasound application. Participants of both groups received a therapeutic ultrasound treatment. Experimental group received first ultrasound and subsequently MEP, while control group was treated only with ultrasound. Ultrasound intervention protocol was performed in the same way for both groups. Application was performed in an adjoining room by another physiotherapist who didn´t know groups. Treatment was carried out with participant in sitting position applying ultrasound at sensitive point marked by examiner of evaluation station. Ultrasound therapy was delivery at 1MHz, 1.5 Watts/cm2, 100% duty cycle (SATP: 1.5Watts/cm2 and SATA:1.5W/cm2), ERA 5cm2 and 15 minutes.24 Once ultrasound intervention was finished, participants of MEP group were taken to microelectrolysis box, while participants of control group returned to evaluation station.
5. Microelectrolysis application. Microelectrolysis was performed by another physiotherapist. Before intervention, puncture area was cleaned with alcohol. Procedure was performed with latex gloves. Acupuncture needle was introduced perpendicular to demarcated point of trapezius with 0.14mA intensity. Dispersing electrode was placed in external surface of contralateral arm once chosen trapezius muscle. Inside tissue intensity was raised to 0.6mA. Each participant was instructed to indicate to physiotherapist appearance of burning, pain or great local pressure in order to pause emission. Emission time was recorded until symptoms appeared, indicating T1 time, pausing emission for 30 seconds. Then a second emission was made until participant referred again discomfort symptoms. Second emission time was recorded as T2, pausing application again for 30 seconds. Third and last emission was delivered for same time obtained for T2 or if discomfort appeared before completing that time.
6. Pain pressure threshold (PPTpre) and pain intensity (PIpre) postintervention evaluation.

Completing intervention, participants returned to evaluation station. Evaluator repeated the same assessment protocol made before ultrasound and MEP application, recording PPT and PI postintervention. Variables PPTdiff1-1 and PIdiff1-1 were created based on differences between algometry and pain intensity measurements before and after intervention. Participants were cited for a reevaluation on day three and seven obtained variables PPT2, PI2, PPT3 and PI3. This allowed to create PPTdiff2-1, PPT3-1, PIdiff2-1 and PIdiff3-1 variables, that represented differences obtained between the measurements of days three and seven with those obtained on day one before intervention.

ELIGIBILITY:
1. Inclusion criteria

   * Students of Sciences Rehabilitation Faculty.
   * Participants over 18 years old.
   * Participants presenting Hypersensitive Pain Points (Trigger Points) at level of upper trapezius muscle. The positive trigger point (+) will be the presence of pain at a pressure of less than 3kg/cm2 at muscle point.
2. Exclusion criteria

   * Musculoskeletal problems or pathologies of the neck or shoulders in the last 6 months (fractures, sprains, tendinopathies, dislocations, muscle tears, etc.).
   * Participants who present cervical pain.
   * Presence of osteosynthesis materials near shoulders, neck or surrounding areas
   * Alterations of sensitivity such as hypesthesia, anesthesia or hyperesthesia in the neck, shoulders and / or arms
   * Presence of wounds or skin alterations in the shoulder region (psoriasis, scars, keloids).
   * Apprehension or fear of electrotherapy aplication.
   * Ingestion of medications or analgesic pharmacological treatment at time of recruitment (Non-steroidal anti-inflammatory or steroidal).
3. Elimination Criteria

   * Non-tolerance of electrotherapy intervention that requires suspension of treatment.
   * Non-completion of evaluation protocol (attendance at all scheduled sessions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hernán A de la Barra Ortiz, Mg., Principal Investigator — Universidad Andrés Bello
Locations (1):
- Universidad Andrés Bello, Santiago, Comuna Las Condes, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleckenstein J, Zaps D, Ruger LJ, Lehmeyer L, Freiberg F, Lang PM, Irnich D. Discrepancy between prevalence and perceived effectiveness of treatment methods in myofascial pain syndrome: results of a cross-sectional, nationwide survey. BMC Musculoskelet Disord. 2010 Feb 11;11:32. doi: 10.1186/1471-2474-11-32. PMID 20149248
- [Background] Currier DP, Mann R. Muscular strength development by electrical stimulation in healthy individuals. Phys Ther. 1983 Jun;63(6):915-21. doi: 10.1093/ptj/63.6.915. PMID 6856678
- [Background] Lewis D, Lewis B, Sturrock RD. Transcutaneous electrical nerve stimulation in osteoarthrosis: a therapeutic alternative? Ann Rheum Dis. 1984 Feb;43(1):47-9. doi: 10.1136/ard.43.1.47. PMID 6364997
- [Background] Kloth LC, Feedar JA. Acceleration of wound healing with high voltage, monophasic, pulsed current. Phys Ther. 1988 Apr;68(4):503-8. doi: 10.1093/ptj/68.4.503. PMID 3258429
- [Background] Mendel FC, Wylegala JA, Fish DR. Influence of high voltage pulsed current on edema formation following impact injury in rats. Phys Ther. 1992 Sep;72(9):668-73. doi: 10.1093/ptj/72.9.668. PMID 1508974
- [Background] Sylvestre JP, Guy RH, Delgado-Charro MB. In vitro optimization of dexamethasone phosphate delivery by iontophoresis. Phys Ther. 2008 Oct;88(10):1177-85. doi: 10.2522/ptj.20080043. Epub 2008 Aug 21. PMID 18719003
- [Background] Conjeevaram R, Banga AK, Zhang L. Electrically modulated transdermal delivery of fentanyl. Pharm Res. 2002 Apr;19(4):440-4. doi: 10.1023/a:1015135426838. PMID 12033377
- [Background] Xia P, Wang X, Lin Q, Cheng K, Li X. Effectiveness of ultrasound therapy for myofascial pain syndrome: a systematic review and meta-analysis. J Pain Res. 2017 Mar 7;10:545-555. doi: 10.2147/JPR.S131482. eCollection 2017. PMID 28331357
- [Background] Lavelle ED, Lavelle W, Smith HS. Myofascial trigger points. Med Clin North Am. 2007 Mar;91(2):229-39. doi: 10.1016/j.mcna.2006.12.004. PMID 17321283
- [Background] Kinser AM, Sands WA, Stone MH. Reliability and validity of a pressure algometer. J Strength Cond Res. 2009 Jan;23(1):312-4. doi: 10.1519/jsc.0b013e31818f051c. PMID 19130648
- [Background] Espejo-Antunez L, Tejeda JF, Albornoz-Cabello M, Rodriguez-Mansilla J, de la Cruz-Torres B, Ribeiro F, Silva AG. Dry needling in the management of myofascial trigger points: A systematic review of randomized controlled trials. Complement Ther Med. 2017 Aug;33:46-57. doi: 10.1016/j.ctim.2017.06.003. Epub 2017 Jun 15. PMID 28735825
- [Background] Wieder DL. Treatment of traumatic myositis ossificans with acetic acid iontophoresis. Phys Ther. 1992 Feb;72(2):133-7. doi: 10.1093/ptj/72.2.133. PMID 1549634
- [Background] Guy RH, Delgado-Charro MB, Kalia YN. Iontophoretic transport across the skin. Skin Pharmacol Appl Skin Physiol. 2001;14 Suppl 1:35-40. doi: 10.1159/000056388. PMID 11509905
- [Background] Kalia YN, Guy RH. The electrical characteristics of human skin in vivo. Pharm Res. 1995 Nov;12(11):1605-13. doi: 10.1023/a:1016228730522. PMID 8592657
- [Background] Uddin Z, MacDermid JC. Quantitative Sensory Testing in Chronic Musculoskeletal Pain. Pain Med. 2016 Sep;17(9):1694-703. doi: 10.1093/pm/pnv105. Epub 2016 Feb 18. PMID 26893116
- [Background] Barbero M, Schneebeli A, Koetsier E, Maino P. Myofascial pain syndrome and trigger points: evaluation and treatment in patients with musculoskeletal pain. Curr Opin Support Palliat Care. 2019 Sep;13(3):270-276. doi: 10.1097/SPC.0000000000000445. PMID 31313700

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group (Ultrasound Therapy): Group treated with conventional ultrasound (US) on MTrP with 1MHz, 1.5W/cm2, 5cm2 ERA, 100% duty cycle and 15 minutes treatment time.
  Ultrasound therapy: Application of conventional ultrasound (US) on PGm with a frequency of treatment 1MHz, intensity of 1.5W / cm2, ERA 5cm2, Duty Cycle 100%, treatment time 6 minutes.
Period: Overall Study
Arm/Group | Percutaneous Microelectrolysis Group (MEP) | Control Group (Ultrasound Therapy)
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Percutaneous Microelectrolysis Group (MEP) | Ultrasound Therapy | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (1.9) | 22.0 (1.6) | 22.3 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 24 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Chile | 24 | 24 | 48
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 24.5 (3.4) | 22.9 (2.3) | 23.6 (2.8)
Short trapezius muscle laterality [Count of Participants; unit: Participants]
  Right | 17 | 20 | 37
  Left | 7 | 4 | 11
SP-AC [Mean (Standard Deviation); unit: centimeters] — Line drawn between C7 spinous process and acromion where the distance from medial to lateral will be marked in which the MTrP will be found.
  centimeters | 9.2 (1.8) | 8.4 (1.7) | 8.7 (1.7)
PPTpre intervention (PPTpre1) [Mean (Standard Deviation); unit: Kg/cm2] | 1.4 (0.2) | 1.4 (0.2) | 1.4 (0.2)
PIpre intervention (PIpre1) [Mean (Standard Deviation); unit: mm] | 32.1 (13.6) | 31.4 (15.1) | 32.0 (14.2)

OUTCOME MEASURES:

1. Primary Outcome: Pain Pressure Threshold (PPT)
Description: Pain Intensity expressed in kilograms per square centimeter(kg/cm2) reported by participants when performing algometry test at sensitive point of upper trapezius muscle. PPT was valued in four occasions: PPT1 pre (baseline), PPT1 post, PPT 2 (at day 3) and PPT 3 (at day 7). PPT will be evaluated through the BASELINE® pressure algometer.
Time Frame: PPTpre1 (baseline), PPTpost1 (post baseline), PPT2 (Day 3), PPT3 (Day 7), assessed an average of 30 minutes at each session
Measure: Mean (Standard Deviation); unit: Kg/cm2
Arm/Group | Percutaneous Microelectrolysis Group (MEP) | Control Group (Ultrasound Therapy)
Number analyzed (Participants) | 24 | 24
Kg/cm2
  PPTpre1 | 1.4 (0.2) | 1.4 (0.2)
  PPTpost1 | 1.6 (0.2) | 1.6 (0.2)
  PPT2 | 1.7 (0.1) | 1.6 (0.2)
  PPT3 | 1.9 (0.3) | 1.7 (0.2)
  PPTdiff1-1 | 0.2 (0.2) | 0.2 (0.1)
  PPTdiff2-1 | 0.4 (0.2) | 0.2 (0.2)
  PPTdiff3-1 | 0.5 (0.4) | 0.3 (0.3)

2. Secondary Outcome: Pain Intensity (PI)
Description: Magnitude of pain expressed in millimeters (mm) referred by participants. PI was evaluated through visual analogue scale at moment of performing pressure algometry test in the sensitive point of upper trapezius muscle. PI was assessed with an analogous visual scale where the participant will mark the pain generated by the algometry on a scale of 1 to 100 millimeters. PI was valued in four occasions: PI1 pre (baseline), PI1 post, PI 2 (at day 3) and PI 3 (at day 7).
Time Frame: PIpre1 (baseline), PIpost1 (post baseline), PI2 (Day 3), PI3 (Day 7), assessed an average of 3 minutes at each session
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Percutaneous Microelectrolysis Group (MEP) | Control Group (Ultrasound Therapy)
Number analyzed (Participants) | 24 | 24
mm
  PIpre1 | 32.1 (13.6) | 31.4 (15.1)
  PIpost1 | 24.6 (12.7) | 24.8 (15.1)
  PI2 | 21.6 (11.0) | 23.8 (14.0)
  PI3 | 18.1 (9.9) | 20.0 (13.2)
  PIdiff1-1 | -7.5 (8.4) | -6.6 (8.6)
  PIdiff2-1 | -10.5 (11.9) | -7.6 (12.1)
  PIdiff3-1 | -14.0 (12.3) | -11.5 (13.1)

ADVERSE EVENTS:
Time Frame: 3 month follow up no adverse events recorded
Description: Not Including adverse event
Arm/Group | Percutaneous Microelectrolysis Group (MEP) | Control Group (Ultrasound Therapy)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
Sample size, determined for convenience. Current dose and number of intervention sessions. Discomfort thresholds were detected at different emission´s times in participants of MEP group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03636386/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03636386/SAP_002.pdf
  • Informed Consent Form (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03636386/ICF_001.pdf